CLINICAL TRIAL: NCT05172531
Title: Efficacy and Safety Profile of Cisatracurium Besylate for Intra-abdominal Hypertensiona: Single Center, Randomized, Controlled Trial
Brief Title: Efficacy and Safety Profile of Cisatracurium Besylate for IAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Department of anesthesiology , Director, Chief physician, Tianjin Nankai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKYY-IAH-2021-12
Record Dates: First submitted 2021-12-27; First posted 2021-12-29 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Intra-abdominal Hypertension
MeSH Terms: conditions — Intra-Abdominal Hypertension | interventions — cisatracurium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Participants in the test group received Cisatracurium Besilate 0.12mg/kg/hr Continuous infusion During intubation
  Interventions: Drug: Cisatracurium Besylate
- control group (Sham Comparator): Participants in the control group received saline 0.12ml/kg/hr Continuous infusion During intubation
  Interventions: Drug: saline 0.12ml/kg/hr

INTERVENTIONS:
Drug: Cisatracurium Besylate — Participants in the test group received Cisatracurium Besylate 0.12mg/kg/hr continuous infusion during intubation。
  Arms: test group
Drug: saline 0.12ml/kg/hr — saline 0.12ml/kg/hr
  Arms: control group

SUMMARY:
This study is a randomized, double-blinded, controlled design. In this study, Cisatracurium Besylate was selected for treatment in Intra-abdominal hypertension or abdominal compartment syndrome,accompanied with evaluating the effects on the duration of organ failure,length of hospital stay and mortality.To clarify the effect of Cisatracurium Besylate on IAH/ACS is of great significance to the clinical applications.

DETAILED DESCRIPTION:
1. Title: Title: Efficacy and Safety Profile of Cisatracurium Besylate on Intra-abdominal hypertension: A Randomized Clinical Trial
2. Research center: single center
3. Design of the research: A randomized, double-blind and parallel controlled study
4. Object of the research: The patients over 18 years that Intra-abdominal pressure over 12mmHg.
5. Sample size of the research: A total of 80patients,40 cases in each group
6. Interventions: Participants in the test group received Cisatracurium Besylate 0.12mg/kg/hr continuous infusion during intubation.while participants in the control group was the same as the test group except for received the same volume of saline instead of Cisatracurium Besylate.TOF-Watch was used to monitor the function of nerve and muscle in two groups and the dose was adjusted according to the TOF value.
7. The aim of the research:To investigate the effect of Cisatracurium Besylate on IIntra-abdominal hypertension or abdominal compartment syndrome.
8. Outcome #Primary outcomes: mortality. Secondary outcomes: Duration of organ failure; Time for enteral nutrition to reach the standard (30kcal/kg); Mechanical ventilation time; Length of hospital stay
9. The estimated duration of the study#1-2years

ELIGIBILITY:
Inclusion Criteria:

1. Intra-abdominal pressure≥12mmHg
2. Age ≥18 years old
3. Obtain informed consent.

Exclusion Criteria:

1. Pregnancy pancreatitis
2. Patients who have undergone percutaneous puncture or surgical drainage before admission, and have undergone surgical decompression due to early abdominal hypertension
3. Patients with a history of chronic organ dysfunction (such as uremia, COPD, liver cirrhosis, heart failure, etc.)
4. Those who refuse to participate in the research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-29 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
All-cause 28-day mortality | 1-2year
  All reasons (such as infection, hemorrhage) caused the mortality during the first 28 days after treatments

SECONDARY OUTCOMES:
Duration of organ failure | an average of 1-2 year
  The time of organ failure recovered
Duration of mechanical ventilation in patients with endotracheal intubation in ICU | an average of 1 year
  Duration of mechanical ventilation in patients with endotracheal intubation in ICU
Length of stay in hospital | 24 months
  ICU stay time and hospitalization time

REFERENCES:
- [Background] Kimball EJ. Intra-abdominal hypertension and abdominal compartment syndrome: a current review. Curr Opin Crit Care. 2021 Apr 1;27(2):164-168. doi: 10.1097/MCC.0000000000000797. PMID 33480617
- [Background] Pereira R, Buglevski M, Perdigoto R, Marcelino P, Saliba F, Blot S, Starkopf J. Intra-abdominal hypertension and abdominal compartment syndrome in the critically ill liver cirrhotic patient-prevalence and clinical outcomes. A multicentric retrospective cohort study in intensive care. PLoS One. 2021 May 13;16(5):e0251498. doi: 10.1371/journal.pone.0251498. eCollection 2021. PMID 33984016
- [Background] De Waele JJ, Benoit D, Hoste E, Colardyn F. A role for muscle relaxation in patients with abdominal compartment syndrome? Intensive Care Med. 2003 Feb;29(2):332. doi: 10.1007/s00134-002-1578-x. No abstract available. PMID 12675044
- [Background] Chiles KT, Feeney CM. Abdominal compartment syndrome successfully treated with neuromuscular blockade. Indian J Anaesth. 2011 Jul;55(4):384-7. doi: 10.4103/0019-5049.84867. PMID 22013257